CLINICAL TRIAL: NCT05022849
Title: A Phase 1, Dose Escalation Study of JNJ-75229414, a Chimeric Antigen Receptor T Cell (CAR-T) Therapy Directed Against KLK2 for Metastatic Castration-Resistant Prostate Cancer
Brief Title: A Study of JNJ-75229414 for Metastatic Castration-resistant Prostate Cancer Participants
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: CR108972; 75229414MPC1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-08-20; First posted 2021-08-26 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1: Dose Escalation (Experimental): Participants will receive a conditioning regimen of cyclophosphamide and fludarabine intravenously (IV) followed by JNJ-75229414 IV infusion escalated sequentially with a targeted dose consistent with the dose required by the cohort being enrolled to determine recommended Phase 2 dose (RP2D) regimen(s). Additional, intermediate dose levels may be implemented based on the review of all available data including, but not limited to, safety, efficacy, pharmacokinetics (PK), and pharmacodynamics (PD) by the study evaluation team (SET). Participants may receive bridging therapy (anti-androgen receptor agents [example, abiraterone, enzalutamide] and radiotherapy, or chemotherapy [example, docetaxel]) if clinically indicated to maintain disease stability.
  Interventions: Drug: JNJ-75229414; Drug: Bridging Therapy
- Part 2: Dose Expansion (Experimental): Participants will receive JNJ-75229414 for each RP2D regimen determined in Part 1.
  Interventions: Drug: JNJ-75229414; Drug: Bridging Therapy

INTERVENTIONS:
Drug: JNJ-75229414 — JNJ-75229414 infusion will be administered intravenously.
  Other Names: KLK2 CAR-T Cells
Drug: Bridging Therapy — Bridging therapy including Anti-AR agents (example, abiraterone, enzalutamide) will be administered orally and radiotherapy, or chemotherapy (example, docetaxel) will be administered intravenously.

SUMMARY:
The purpose of this study is to determine recommended Phase 2 dose (RP2D) regimen(s) of JNJ-75229414 in Part 1 (Dose Escalation and to determine safety at the RP2D regimen(s) in Part 2 (Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

* Histology: Metastatic CRPC (mCRPC) with histologic confirmation of adenocarcinoma. Metastatic CRPC with neuroendocrine features or mixed histology is excluded
* Prior Therapy: Prior treatment with at least 1 prior novel androgen receptor AR-targeted therapy (that is, abiraterone acetate, apalutamide, enzalutamide, darolutamide), or at least 1 prior chemotherapy (example, docetaxel)
* Eastern Cooperative Oncology Group (ECOG) Performance Status grade of 0 or 1
* Measurable disease by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 or detectable prostate-specific antigen (PSA) levels based on local laboratory results
* Fertile participants must use a condom with spermicide during any sexual contact with a woman of childbearing potential, including pregnant women, from the time of signing the ICF until 1 year after receiving a JNJ-75229414 infusion. Vasectomized participants must agree to use a condom to protect any sexual partner from exposure to semen for 1 year after receiving the last dose of study drug. Contraceptive (birth control) use should be consistent with local regulations regarding the acceptable methods of contraception for those participating in clinical studies

Exclusion Criteria:

* Prior Grade 4 Cytokine release syndrome (CRS) or Grade 3 or Grade 4 neurotoxicity related to any T cell redirection (Bispecific cluster of differentiation [CD 3])
* Prior Kallikrein 2 (KLK2)-targeted therapy
* Prior chimeric antigen receptor T cell (CAR-T) therapy
* Receiving systemic treatment less than or equal to (<=) 6 months prior to signing informed consent) for any invasive malignancy other than prostate cancer unless approved by the sponsor. Bisphosphonates initiated greater than or equal to (>=) 6 weeks prior signing informed consent are allowed
* Less than 2 weeks between last administration anti-androgen agents (example, abiraterone or enzalutamide), poly adenosine diphosphate-ribose polymerase (PARP) inhibitors (example, olaparib) or radiotherapy, and less than 3 weeks between last administration of cytotoxic chemotherapy (example, docetaxel), radionuclides (example, radium-223, lutetium-177-Prostate-specific membrane antigen [PSMA]-617) or an investigational agent, and apheresis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-09-28 (Actual); Primary Completion 2037-10-30 (Estimated); Study Completion 2037-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 15 years 9 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Number of Participants with AEs by Severity | Up to 15 years 9 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event.
Part 1: Number of Participants with Dose-limiting Toxicity (DLT) | Up to 28 days
  Number of participants with DLT will be assessed. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Maximum Observe Plasma Concentration (Cmax) of JNJ-75229414 | Up to 15 years 9 months
  Cmax is the maximum observed plasma concentration of JNJ-75229414.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of JNJ-75229414 | Up to 15 years 9 months
  Tmax is the actual sampling time to reach maximum observed plasma concentration of JNJ-75229414.
Area Under Plasma Concentration Versus Time Curve from Time Zero to t Time (AUC[0-t]) of JNJ-75229414 | Up to 15 years 9 months
  AUC(0-t) is the area under the plasma concentration versus time curve from time zero to 't' time.
Peripheral T Cell Expansion and Persistence via Monitoring Chimeric Antigen Receptor T (CAR-T) Positive Cell Counts | Up to 15 years 9 months
  Peripheral T cell expansion and persistence via monitoring CAR-T positive cell counts will be reported.
Number of Participants With Presence of Anti-JNJ-75229414 Antibodies | Up to 15 years 9 months
  Number of participants with antibodies to JNJ-75229414 will be reported.
Overall Response Rate (ORR) | Up to 15 years 9 months
  ORR is defined as the percentage of participants who achieve a confirmed best overall response of Complete Response (CR) or Partial Response (PR) evaluated by an independent local radiology review based on Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Prostate Cancer Working Group 3 (PCWG3) criteria will be used to assess progressive bone metastases.
Disease Control Rate (DCR) | Up to 15 years 9 months
  DCR is defined as the sum of CR, PR, and stable disease (SD).
Duration of Response (DoR) | Up to 15 years 9 months
  DoR is defined as the time from the date of first documented responses until date of documented progression or death whichever comes first.
Time to response (TTR) | Up to 15 years 9 months
  TTR defined as the time from the date of first dose of study drug to the date of first documented response.
Peripheral Blood Quantitation of Vesicular Stomatitis Virus G glycoprotein (VSV-G) Copy Numbers | Up to 15 years 9 months
  Peripheral blood quantitation of VSV-G copy numbers will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (8):
- United States (8):
  - City of Hope Cancer Center, Duarte, California
  - Norton Cancer Institute, Louisville, Kentucky
  - University Of Minnesota, Minneapolis, Minnesota
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Utah Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency